CLINICAL TRIAL: NCT01353456
Title: Multimodal Analgesic Using Morphine and COX-2 With or Without Dexmedetomidine for Colorectal Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Cheung Chi Wai, Clinical Associate Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 200907176018
Record Dates: First submitted 2011-05-04; First posted 2011-05-13 (Estimated); Last update posted 2013-04-04 (Estimated); Status verified 2013-04

CONDITIONS: Pain, Postoperative
Keywords: Ambulation; Side effects; Serum sCD40L; Bowel function; Postoperative pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Dexmedetomidine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dexmedetomidine (Active Comparator)
  Interventions: Drug: Dexmedetomidine
- Normal saline (Placebo Comparator)
  Interventions: Drug: Normal Saline

INTERVENTIONS:
Drug: Dexmedetomidine — Patient will receive a loading dose of 1μg/kg (0.25ml/kg) intravenous dexmedetomidine over 10 minutes before induction, and then followed by continuous infusion at a rate of 0.5μg/kg/h (0.125ml/kg/h) until wound closure.
  Arms: Dexmedetomidine
Drug: Normal Saline — Same volume as dexmedetomidine given
  Arms: Normal saline

SUMMARY:
Recently, multimodal approach for postoperative pain control has been advocated.Combinations of traditional and novel pharmacological agents are administered, aiming to improve analgesia, spare opioid consumption, minimise adverse effects, and improve postoperative bowel function in colorectal surgery.

One of the novel agents suggested is dexmedetomidine. It is a selective alpha-2 adrenoceptor agonist, which has been demonstrated to have anaesthetic, sedative and analgesic-sparing effects. Furthermore, a significant reduction in postoperative morphine consumption by using patient-controlled analgesia (PCA) has been achieved when dexmedetomidine was administered before operation. The drug also reduces cate-cholamine secretion, thereby reducing stress and leading to a modest reduction in heart rate and blood pressure, which may be particularly beneficial in patients with cardiovascular disease, while respiratory rate is not affected.

In this study, the investigators would like to evaluate the analgesic effects of dexmedetomidine, which is administered intraoperatively with morphine, followed by postoperative PCA morphine infusion, for postoperative pain for open and laparoscopic colorectal surgery. Cyclooxy-genase-2 (COX-2) inhibitors and rescue intramuscular pethidine will also be incorporated as part of the multimodal analgesia regimens.

Good pain control can help to decrease cardiovascular complications. Emerging data has suggested a key role of soluble CD40L as inflammatory mediators of atherosclerotic lesion progression. The investigators would like to evaluate the effect of our analgesic regimens on soluble CD40L peri-operatively.

The investigators hypothesize that intraoperative dexmedetomidine can reduce postoperative pain and improve recovery and outcomes.

DETAILED DESCRIPTION:
PROCEDURES:

Patients will be approached at the pre-admission clinic or in the general ward before operation. The analgesic modalities will be explained and patient will be recruited into study if s/he agrees. Patient will then be randomised into one of the two groups receiving intraoperative morphine with dexmedetomidine then postoperative PCA morphine (D), or intraoperative morphine only then postoperative PCA morphine (M).

Randomisation, blinding, and preparation of dexmedetomidine and placebo Patients who undergo open and laparoscopic colonic and rectal surgery will be stratified in randomisation. For each type of operation (colonic and rectal), randomisation will be based on using blocks of 5 patients to ensure both groups having equal sample size. A computer-generated random sequence will be used to select the allocation order.

Both patients and investigators will be blinded to the allocated analgesic modalities, i.e. the administration of dexmedetomidine. Dexmedetomidine or normal saline (placebo) will be prepared by clinical staff who will not participate in observation and data analysis.

For group D, dexmedetomidine will be prepared by adding 2ml of the drug (100μg/ml) to 48ml of 0.9% sodium chloride injection, which make up to a total of 50ml. The final concentration for administration is thus 200μg in 50ml, i.e. 4μg/ml.

For group M, a syringe of 50ml normal saline will be prepared as placebo. As both dexmedetomidine and placebo will look the same as 50ml clear liquid in syringe, both patient and investigator will be blinded to the substance administered.

Preoperative care:

The patients will be assessed at pre-admission clinic or at the general ward. Blood for soluble CD40L with other routine investigations will be taken. Bowel preparation will start one day before operation. Patient will fast since midnight before operation.

Anaesthesia and intraoperative care:

Both groups of patients will be anaesthetised according to the protocol as follow:

Patient will receive no sedative premedication. On arrival in the operation theatre, a 16-gauge intravenous cannula will be placed under local analgesic. Pulse, pulse oximetry and non-invasive blood pressure measurement will be checked every 5 minutes throughout the operation.

Propofol 2mg/kg, fentanyl 1.5μg/kg and atracurium 0.5mg/kg will be used for general anaesthesia induction. Anaesthesia will be maintained with mixture of isoflurane, air and oxygen. Isoflurane concentration will be titrated to optimal heart rate and blood pressure by the anaesthesiologist.

Thermal blanket and infusion fluid warmer will be used to aim at maintaining core body temperature at 35.5 to 37.5 degrees Celsius. A urinary catheter will be inserted to monitor urine output. Intermittent pneumatic compression device will be applied to the lower limbs for deep vein thrombosis prophylaxis.

At the discretion of the anaesthesiologist, hypotension will be treated with intravenous ephedrine or phenylephrine. Hypertension or tachycardia will be treated with isoflurane up to 2% end-tidal concentration (~1.5 MAC). If persisted, beta-blockers such as labetalol or arterial vasodilators such as hydralazine may be given.

Isoflurane will be switched off after closure of the inner layer of the wounds. Reversal will be achieved by intravenous neostigmine 50μg/kg and atropine 20μg/kg after operation. Patient will then be transferred to recovery room for monitoring for at least 1 hour.

Analgesic modalities and pain assessment:

Procedures for the two analgesic modalities are described below:

Group D: intraoperative morphine with dexmedetomidine then postoperative PCA morphine. Patient will receive a loading dose of 1μg/kg (0.25ml/kg) intravenous dex-medetomidine over 10 minutes before induction, and then followed by continuous infusion at a rate of 0.5μg/kg/h (0.125ml/kg/h) until wound closure. Bolus dose of 0.1mg/kg morphine sulphate will be given intravenously prior to incision. At the third and forth hour, morphine sulphate 0.1mg/kg may be given in divided dose titrated to patient's response. On arrival in the recovery room, boluses of 2mg intravenous morphine will be given every 5 minutes until NRS pain score is less than 4. A PCA machine will then be connected. The machine will be configured to give 1mg of morphine at a time and the lockout duration will be set to 5 minutes. No basal infusion will be given and the maximum dose limit will be 0.1mg/kg per hour.

Group M: intraoperative morphine then postoperative PCA morphine. All procedures for Group D patients will be followed, but dexmedetomidine administration will be replaced by placebo (normal saline) of the same volume and rate.

Both groups: Starting from postoperative day 1, when patient resumes fluid diet, oral celecoxib 200mg will be given twice daily for 3 days or until discharge, whichever earlier. From day 4 onwards, one tablet of dologesic (paracetamol plus dextropropoxyphene) will be given every 4 hours as needed until discharge.

From postoperative day 0, rescue analgesic in the form of intramuscular pethidine 0.5mg/kg will be prescribed every 4 hours if necessary.

During the administration of PCA morphine, respiratory rate, SpO2 and sedation score will be monitored every hour; blood pressure and pulse, numerical rating scale (NRS) pain scores at rest and during cough, cumulative doses and tries/goods, as well as side effects will be recorded every 4 hours. Patient will be seen by anaesthesiologist every day to assess the adequacy of analgesia.

PCA morphine will be administered for at least 2 days. On postoperative day 2, if NRS pain scores during cough is less than 4 on a clinically low morphine consumption, PCA will be stopped; if equals or greater than 4, or still on a high PCA consumption, it will be continued. Assessment will be repeated daily. If NRS pain score during cough remains at 4 or above on day 5, patient will be evaluated for complications and managed at the discretion of the anaesthesiologist.

After PCA morphine has stopped, NRS pain scores at rest and during cough, dose and frequency of rescue analgesia used will be charted once a day until discharge.

Postoperative care and assessment:

Early mobilisation is encouraged after operation. On postoperative day 1, patient will be put on fluid diet.

The surgical team will be responsible for postoperative assessments, such as recording daily gastrointestinal function (bowel sound, flatus and bowel opening), postoperative complications (if any) and readiness for discharging patient (good pain control with oral analgesics, ambulatory, resumption of bowel function, i.e. stool or flatus, have 2 to 3 feeds without vomiting or abdominal distension).

Blood for soluble CD40L and other routine investigations will be taken at post-operative day 2.

Patient's satisfaction on analgesia will be asked using NRS from zero to 10 upon discharge.

DATA COLLECTION:

The following data will be collected:

* Demographics
* Time of admission
* Type of colorectal surgery and incision
* Intraoperative vital signs (blood pressure, pulse, pulse oximetry)
* Estimated intraoperative blood loss
* Volume of intraoperative fluid/blood infusion
* Duration of anaesthetic/analgesic procedures before surgical procedures
* Duration of surgical procedures
* Time from end of surgical procedures to extubation
* Tries and goods of PCA use
* Cumulative morphine consumption
* NRS pain scores at rest and during cough and vital signs upon recovery, hourly for 4 hours, then 4-hourly during PCA morphine up to 5 days, and daily afterwards until discharge
* Dose and frequency of rescues analgesic (IM pethidine) use
* Side effects of analgesics, if any (pruritis, dizziness, nausea, vomiting, etc.)
* Time to recovery of bowel functions (bowel sound, flatus and bowel opening)
* Time to recovery of food intake (fluid, semisolid and solid diet)
* Time to ambulation (bed rest, sit up, sit out of bed, walk with aid, walk without aid)
* Surgical and anaesthetic complications, if any (ileus, perineal abscess, wound infection, urinary retention, etc.)
* Time to discharge
* Patient's satisfaction upon discharge
* Persistent pain 6 months after operation
* Survival status 6 and 12 months after operation
* Soluble CD40L preoperatively and at post-operative day 2 If, at certain time point after operation, patient is unable to be managed according to protocol due to any reason such as development of complication, no further data will be collected.

DATA ANALYSIS:

The intention-to-treat principle will be used. In other words, patient will be included and remained in their designated groups for data analysis even if there is a change in surgical or anaesthetic/analgesic management, as long as they have had an open or laparoscopic abdominal incision during operation.

Statistical methods used:

* Intraoperative vital signs, estimated blood loss, duration of anaesthetic/analgesic and surgical procedures, time to extubation, tries and goods of PCA use, cumulative morphine consumption, dose and frequency of rescue analgesic use, time to recovery of bowel functions, food intake and ambulation, time to discharge: Student's t-test
* NRS pain scores, patient's satisfaction: Mann-Whitney U test
* Side effects and postoperative complications: binary logistic regression

ELIGIBILITY:
Inclusion Criteria:

* ASA I to III
* Age 18 to 80 years
* Scheduled for elective open and laparoscopic colonic or upper rectal resection in Queen Mary Hospital in Hong Kong

Exclusion Criteria:

* Extended resection involving other organs such as liver and urinary bladder
* Known drug allergy to alpha-2 agonists, opioids, non-steroidal anti-inflammatory drugs (NSAIDs) including COX-2 inhibitors or sulphonamides
* Regular use of clonidine, methyldopa, opioids or psychiatric drugs
* Alcohol or drug abuse
* Known history of second or third degree heart block, ischaemic heart disease, valvular heart disease, or heart failure
* Known history of pulmonary embolism or deep vein thrombosis
* Known history of sleep apnoea syndrome
* Impaired renal function, defined as preoperative serum creatinine level over 120µmol/L
* Impaired hepatic function, defined as preoperative serum albumin level less than 30g/L
* Impaired or retarded mental state
* Not self-ambulatory before operation
* Difficulties in using patient-controlled analgesia
* BMI > 35kg/m2
* Pregnancy
* Patient refusal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2008-05; Primary Completion 2010-03 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Postoperative pain score as Numerical Rating Scale | 5 days

SECONDARY OUTCOMES:
Number of patients having flatus and blow opening | 5 days
Serum level of sCD40L | 3 days

CONTACTS AND LOCATIONS:
Locations (1):
- Queen Mary Hosspital, Hong Kong, China